CLINICAL TRIAL: NCT01351259
Title: Continuous Control of Polyurethane Tracheal-cuff Pressure: Efficiency of a Pneumatic Device
Acronym: Nosten
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Principal Investigator, Saad NSEIR, Dr, University Hospital, Lille
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-A00598-49; 2009_20/0925 (Other: sponsor)
Record Dates: First submitted 2011-05-09; First posted 2011-05-10 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-08

CONDITIONS: Mechanical Ventilation Complication; Tracheal Intubation Morbidity
Keywords: Mechanical ventilation; Intubation; Cuff pressure; Microaspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Pneumatic device, tapered cuff (Experimental): Intervention: continuous control of cuff pressure using a pneumatic device, tapered polyurethane cuff
  Interventions: Device: Pneumatic device, cylindrical or tapered cuff
- Pneumatic device, cylindrical cuff (Experimental): Continuous control of cuff pressure using a pneumatic device in patients intubated with cylindrical polyurethane cuffed tracheal tubes
  Interventions: Device: Pneumatic device, cylindrical or tapered cuff
- Routine care, tapered cuff (Active Comparator): Routine care of cuff pressure using a manometer, tapered polyurethane cuff
  Interventions: Device: Pneumatic device, cylindrical or tapered cuff
- Routine care, cylindrical cuff (Active Comparator): Routine care of cuff pressure using a manometer, cylindrical polyurethane tracheal cuff
  Interventions: Device: Pneumatic device, cylindrical or tapered cuff

INTERVENTIONS:
Device: Pneumatic device, cylindrical or tapered cuff — Continuous control of cuff pressure using a pneumatic device (Nosten) Cylindrical (Kimberly Clark tube) or tapered (Covidien tube) tracheal cuff
  Other Names: Nosten; Kimberly clark; Covidien

SUMMARY:
Underinflation and overinflation of tracheal cuff are common in intubated patients, including those intubated with polyurethane-cuffed tubes. The aim of this study is to determine the efficiency of a pneumatic device in controlling cuff pressure.

DETAILED DESCRIPTION:
Underinflation and overinflation of tracheal cuff are associated with severe complications such as microaspiration of contaminated secretions, and tracheal ischemia. Efficient control of cuff pressure would probably allow reducing complications related to variations in cuff pressure.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring intubation in the ICU
* Predicted duration of mechanical ventilation > or = 48h
* Age > or = 18 years

Exclusion Criteria:

* Contraindication for semirecumbent position
* Contraindication for enteral nutrition
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2010-02; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with underinflation or overinflation of cuff pressure | 48 h
  Continuous recording of cuff pressure will be performed during 2 24-h periods (with or without the pneumatic device)

SECONDARY OUTCOMES:
Impact of tracheal-cuff shape on variations in cuff pressure | 48 h
  Patients will be intubated with cylindrical or tapered polyurethane cuffed tubes.
Impact of continuous control of cuff pressure on microaspiration of gastric contents | 48 h
  Pepsin will be quantitatively measured in tracheal aspirates of all patients during the 2 24-h periods (with or without the pneumatic device)
Impact of tracheal cuff shape on microaspiration of gastric contents | 48 h
  Pepsin level in tracheal aspirates will be compared between patients intubated with cylindrical polyurethane cuffed-tubes versus those intubated with tapered polyurethane cuffed-tubes

CONTACTS AND LOCATIONS:
Overall Officials: Saad NSEIR, MD, Principal Investigator — CHU de Lille
Locations (1):
- ICU, Calmette Hospital, CHU de Lille, Lille, Nord, France

REFERENCES:
- [Derived] Jaillette E, Zerimech F, De Jonckheere J, Makris D, Balduyck M, Durocher A, Duhamel A, Nseir S. Efficiency of a pneumatic device in controlling cuff pressure of polyurethane-cuffed tracheal tubes: a randomized controlled study. BMC Anesthesiol. 2013 Dec 26;13(1):50. doi: 10.1186/1471-2253-13-50. PMID 24369057